CLINICAL TRIAL: NCT02962570
Title: Comparison of an On-Demand Oxygen Delivery System to Continuous Flow Supplemental Oxygen in the Operating/Procedure Room
Brief Title: On-Demand Oxygen Delivery System Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kai Kuck, Ph.D., University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00094640
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Oxygen Delivery; Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Only Arm (Experimental): Two minutes: Intervention: Device: On Demand Oxygen Delivery 20 sec or 3 breaths, whatever comes first: Intervention: Device: Oxygen Flow Stopped
  Two minutes intervention: Device: Traditional, Always-On, Oxygen Delivery 20 sec or 3 breaths, whatever comes first: Intervention: Device: Oxygen Flow Stopped
  Repeat until the end of the surgical procedure
  Interventions: Device: On Demand Oxygen Delivery; Device: Traditional, Always-On, Oxygen Delivery; Device: Oxygen Flow Stopped

INTERVENTIONS:
Device: On Demand Oxygen Delivery — Supplemental oxygen flow is controlled such that it is on only during inhalation.
Device: Traditional, Always-On, Oxygen Delivery — Supplemental oxygen flow is constantly on, irrespective of whether the patient is inhaling or exhaling.
Device: Oxygen Flow Stopped — Supplemental oxygen flow is stopped completely for a brief period to allow undisturbed end-tidal oxygen and CO2 measurements

SUMMARY:
The main goal of this study is to determine if supplemental oxygen given only when the patient is inspiring (demand delivery) is more effective than constant-flow oxygen given during all phases of the breath regardless if the patient is breathing it in. A previous study in volunteers (NCT02886312) showed that the oxygen saturation in the blood and the concentration of oxygen breathed out from the lungs (end-tidal oxygen) was higher when given in demand (inhalation only) mode. A secondary goal is to determine in patients, whether turning oxygen delivery off during expiration improves the accuracy of end-tidal CO2 (Carbon Dioxide) monitoring. This was found to be the case in the previous volunteer study.

The investigators want to determine if these improvements are also observable in relatively healthy patients undergoing procedural sedation and analgesia. The efficacy of the demand mode will be determined by measuring the resulting difference in oxygen saturation and end-tidal oxygen levels. The investigators will alternate between traditional oxygen delivery (continuous flow) and demand delivery (flow only during inhalation) for two minutes in each mode after which oxygen saturation and end-tidal oxygen will be measured. End-tidal CO2 measurement will be compared with those during the brief time when O2 flow is stopped.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-III

Exclusion Criteria:

* Procedures scheduled for a lime less than 20 minutes
* Age < 18 years
* Baseline SpO2 (arterial oxygen saturation as measured by pulse oximetry) < 93% on room air
* ARDS (Acute respiratory distress syndrome), lung disease, cardiovascular disease
* ASA class IV or above
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
End-tidal Oxygen | measured every 140 seconds minutes throughout the surgical procedure
  Did the novel system increase end-tidal oxygen?
Oxygen Saturation | measured continuously with every heart beat (i.e., approx. every 500-2000msec) throughout the surgical procedure
  Did the novel system increase oxygen saturation?
End-tidal Carbon Dioxide | measured every 140 seconds minutes throughout the surgical procedure
  Was end-tidal carbon dioxide measured more accurately using the novel system?

CONTACTS AND LOCATIONS:
Overall Officials: Kai Kuck, Ph.D., Principal Investigator — University of Utah Department of Anesthesiology
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Bliss PL, McCoy RW, Adams AB. Characteristics of demand oxygen delivery systems: maximum output and setting recommendations. Respir Care. 2004 Feb;49(2):160-5. PMID 14744265
- [Background] Fuhrman C, Chouaid C, Herigault R, Housset B, Adnot S. Comparison of four demand oxygen delivery systems at rest and during exercise for chronic obstructive pulmonary disease. Respir Med. 2004 Oct;98(10):938-44. doi: 10.1016/j.rmed.2004.03.010. PMID 15481269
- [Background] Godbold S, Lowe G, Willis R. Healthcare Professionals Accuracy and Consistency in Setting Oxygen Flowmeters for Patients in an Intensive Care Unit. Respir. Care 59(10):OF26, December 2014.